CLINICAL TRIAL: NCT02145416
Title: Anal Squamous Cell Carcinoma: Investigation of Functional Imaging During chemoRadioTherapy
Brief Title: ART: Anal Squamous Cell Carcinoma: Investigation of Functional Imaging During chemoRadioTherapy
Acronym: ART
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: OCTO-051
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Anal Cancer
Keywords: Imaging; Chemoradiotherapy
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a single arm, single centre imaging study which will be offered to all consecutive, eligible patients receiving radical chemoradiation therapy (CRT) for anal cancer within Oxford University Hospitals.

Investigations

* Dynamic contrast enhanced magnetic resonance imaging (DCE MRI)
* Diffusion weighted magnetic resonance imaging (DWI MRI)
* MRI scan designed to measure the T1 or produce T1-weighed images (T1 MRI)
* MRI scan designed to measure the T2* or produce T2*-weighed images (T2* MRI)
* Perfusion computed tomography (pCT)
* Fludeoxyglucose positron emission tomography (FDG PET/CT)

Study Design: Observational

Target Population: Patients undergoing radical CRT for anal cancer in Oxford University Hospitals National Health Service (NHS) Trust.

Duration on study: Patients should be on study for a maximum of 5 months.

Patient care post-trial: Follow up as per local standard.

No. of Study Site(s): Single Centre, United Kingdon (UK)

End of study: Last Patient, last assessment of response. Patients should be on study for a maximum of 5 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive primary squamous carcinoma of the anus.
* Patients must be fit and scheduled to receive radical CRT with curative intent.
* Any stage tumor 2-node 0 (T2N0)
* Male or female, Age 18 years+.
* The patient is willing and able to comply with the images and protocol for the duration of the study.
* Written (signed and dated) informed consent.

Exclusion Criteria:

* Pregnant or breast-feeding women or women of childbearing potential unless effective methods of contraception are used.
* Previous pelvic radiotherapy
* Patients with a pacemaker or any other implanted metal which would preclude MRI scan.
* Patients with a prosthetic hip.
* Patients receiving radiotherapy with palliative intent.
* Active medical or psychological illness that would render the patient unsuitable for the additional imaging proposed in this study, at the discretion of the investigator

Additional criteria for optional oxygen breathing procedure:

* Patients with Chronic Obstructive Pulmonary Disease
* Any patient not felt to be suitable for supplementary oxygen as considered by an appropriately trained clinician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients receiving radical CRT for anal cancer within Oxford University Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2015-01-27 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2018-04-12 (Actual)

PRIMARY OUTCOMES:
Changes on DW MRI during CRT in anal cancer. | Fraction 8-10 of CRT (Day 10-12) compared with prior to CRT (Day 1)
  The number of patients with a change in ADC values of <20% between pre-CRT DW MRI and repeat DW MRI following 8-10 fractions of CRT

SECONDARY OUTCOMES:
Changes on DCE MRI, Perfusion CT, T2* MRI, FDG PET | Fraction 8-10 of CRT (Day 10-12)
  Changes on alternative functional imaging modalities following 8-10 fractions of CRT:
  * DCE MRI - Change in amplitude and rate of gadolinium enhancement.
  * Perfusion CT - Changes in perfusion maps represented by blood flow, blood volume, mean transition time and permeability surface area.
  * T2* MRI - Change in T2* values in hypoxic regions (with or without oxygen)
  * FDG PET - Change in tumour uptake (% change in SUVmax).
Correlation of findings on different functional images. | Both prior to CRT day 1 and fraction 8-10
  Correlate size and position of regions of poor vascularity / hypoxia between different images at the same timepoint using volume, centre of mass and overlap comparisons.
Correlation of baseline functional images with outcome of CRT | 3 months post CRT compared with prior to CRT (Day 1)
  Compare volumes of poor vascularity / hypoxia in baseline scans (as described above) with complete response rates 3 months after CRT.
Correlation of the change in functional images over CRT with outcome of CRT | 3 months post CRT
  Change in volumes of poor vascularity / hypoxia in baseline scans (as described above) with complete response rates 3 months after CRT.

OTHER OUTCOMES:
Evaluate the use of T1 mapping in anal cancer | Fraction 8-10 of CRT (Day 10-12)
  Evaluate change in T1 value (with or without oxygen) and compare with other MRI images.
Evaluate use of dynamic data acquired during FDG PET scan | Prior to CRT day 1 and Fraction 8-10 (Day 10-12)
  Analyse baseline data from FDG PET scans at baseline and 8-10 fractions of CRT and compare to static scan results.
To use PET SUV data in a radiotherapy in silico modelling exercise to determine if dose sparing of active pelvic bone marrow (PBM) is possible without compromising target coverage by radiation. | Prior to CRT day 1, Fraction 8-10 (Day 10-12) and at end of CRT
  Compare active PBM regions at baseline and Fraction 8-10 on FDG-PET scans to identify regions of RT induced suppression of active PBM Correlate suppressed active PBM regions with dose received and determine if radiotherapy re-planning could spare active regions without compromising target coverage or sparing of organs at risk (OARs).

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Muirhead, MBCHB, MRCP, FRCR, MD, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- Churchill Hospital, Oxford, United Kingdom

REFERENCES:
- [Derived] Robinson M, Muirhead R, Jacobs C, Cooke R, Chu KY, Van den Heuvel F, Ng S, Virdee P, Strauss V, Hawkins M. Response of FDG avid pelvic bone marrow to concurrent chemoradiation for anal cancer. Radiother Oncol. 2020 Feb;143:19-23. doi: 10.1016/j.radonc.2019.08.016. Epub 2019 Sep 7. PMID 31506182
- [Derived] Sabbagh A, Jacobs C, Cooke R, Chu KY, Ng SM, Strauss VY, Virdee PS, Hawkins MA, Aznar MC, Muirhead R. Is There a Role for an 18F-fluorodeoxyglucose-derived Biological Boost in Squamous Cell Anal Cancer? Clin Oncol (R Coll Radiol). 2019 Feb;31(2):72-80. doi: 10.1016/j.clon.2018.11.034. Epub 2018 Dec 21. PMID 30583927